CLINICAL TRIAL: NCT02254473
Title: Evaluating the Efficacy of Lateral Heel Wedges of Osteoarthritis of the Knee
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment.
Sponsor: HealthPartners Institute (Other)
Collaborators: University of Minnesota (Other); Minnesota Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1405M50501
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Results first posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2017-02

CONDITIONS: Knee Osteoarthritis
Keywords: Knee; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wedge Insert (Experimental): Patients will receive a wedge insert
  Interventions: Other: Wedge Insert
- Flat insert (Placebo Comparator): Patients will receive a flat insert
  Interventions: Other: Flat Insert

INTERVENTIONS:
Other: Wedge Insert
  Arms: Wedge Insert
Other: Flat Insert
  Arms: Flat insert

SUMMARY:
This study is looking at the efficacy of a sloped insole in patients with knee osteoarthritis. Regularly wearing a sloped insole over the course of one year will result in a wider joint space by x-ray in 60% of the subjects, a significant decrease in knee pain, decreased use of over the counter analgesics, and a clinically important improvement in the Womac pain and stiffness scale.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 30 years or older with medial compartment knee Osteoarthritis (unilateral) and Grade 4 Kellgren-Lawrence39 radiographic changes presenting for treatment of knee pain.
* Range of motion knee-flexion beyond 100 degrees and not lacking more than 15 degrees of extension.
* Subtalar and forefoot motion permitting foot/ankle eversion with weight bearing.
* Sufficient shoe toe box height to allow space for the insole and therefore comfort and compliance.
* Passive laxity of medial capsule and collateral ligament by knee extension test.

Exclusion Criteria:

* All other forms of knee arthritis other than OA.
* Knee Instability- medial pseudo-opening of greater than grade 1 or detectable Anterior-posterior instability.
* Less than Grade 4 Kellgren-Lawrence radiographic changes in the medial compartment of the knee39.
* Grade 2 or greater Kellgren-Lawrence radiographic39 involvement of the patellofemoral or lateral compartment.
* Inadequate knee range of motion
* Balance problems requiring the use of a walker or wheel chair - ambulation with aid
* Diabetics with peripheral neuropathy
* Knee surgery within the past year
* Intraarticular steroid injection or visco supplementation within 6 months
* Stiff subtalar or forefoot joints - clinical test
* Inadequate shoe toe box depth to accommodate the test or control inserts
* Charcot joint
* Fixed contracture of the medial capsule and/or collateral ligament- clinical test

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-08; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- TRIA Orthopaedic Center, Bloomington, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Wedge Insert: Patients will receive a wedge insert
  Wedge Insert
- Flat Insert: Patients will receive a flat insert
  Flat Insert
Period: Overall Study
Arm/Group | Wedge Insert | Flat Insert
Started | 9 | 3
Completed | 7 | 2
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wedge Insert | Flat Insert | Total
Number analyzed (Participants) | 9 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 0 | 5
  >=65 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 3 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Function and Pain
Description: Tegner: Tegner activity level scale is a graduated list of activities of daily living, recreation, and competitive sports. The scale is 0 to 10 where 10 corresponds to normal function and 0 to unable to perform.
Time Frame: Baseline
Measure: Mean (Full Range); unit: score on a scale 0-10 (normal)
Arm/Group | Wedge Insert | Flat Insert
Number analyzed (Participants) | 9 | 3
score on a scale 0-10 (normal) | 3.66 [1 to 6] | 4.66 [4 to 5]

2. Primary Outcome: Patient Reported Function and Pain
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Full Range); unit: score on a scale 0-10 (normal)
Arm/Group | Wedge Insert | Flat Insert
Number analyzed (Participants) | 9 | 3
score on a scale 0-10 (normal) | 3.77 [1 to 6] | 4 [2 to 5]

3. Primary Outcome: Patient Reported Function and Pain
Description: as for outcome 1
Time Frame: 3 months
Measure: Mean (Full Range); unit: score on a scale 0-10 (normal)
Arm/Group | Wedge Insert | Flat Insert
Number analyzed (Participants) | 8 | 3
score on a scale 0-10 (normal) | 3.88 [1 to 7] | 3.66 [2 to 5]

4. Primary Outcome: Patient Reported Function and Pain
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (Full Range); unit: score on a scale 0-10 (normal)
Arm/Group | Wedge Insert | Flat Insert
Number analyzed (Participants) | 6 | 2
score on a scale 0-10 (normal) | 3.66 [1 to 6] | 3.5 [2 to 5]

5. Primary Outcome: Patient Reported Function and Pain
Description: as for outcome 1
Time Frame: 9 months
Measure: Mean (Full Range); unit: score on a scale 0-10 (normal)
Arm/Group | Wedge Insert | Flat Insert
Number analyzed (Participants) | 8 | 2
score on a scale 0-10 (normal) | 3.88 [1 to 7] | 4 [3 to 5]

6. Primary Outcome: Patient Reported Function and Pain
Description: as for outcome 1
Time Frame: 12 months
Measure: Mean (Full Range); unit: score on a scale 0-10 (normal)
Arm/Group | Wedge Insert | Flat Insert
Number analyzed (Participants) | 6 | 2
score on a scale 0-10 (normal) | 3.17 [1 to 6] | 4 [3 to 5]

7. Secondary Outcome: Kellgren and Lawrence Classification of Osteoarthritis of Knee
Description: X-Ray used to measure Kellgren and Lawrence Classification of Osteoarthritis of Knee (joint space in the knee).
Time Frame: Baseline
Population: Data was not gathered due to pre-mature termination of the study.
Arm/Group | Wedge Insert | Flat Insert
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Kellgren and Lawrence Classification of Osteoarthritis of Knee
Description: X-Ray used to measure Kellgren and Lawrence Classification of Osteoarthritis of Knee (joint space in the knee).
Time Frame: 6 months
Population: Data was not gathered due to pre-mature termination of the study.
Arm/Group | Wedge Insert | Flat Insert
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Wedge Insert | Flat Insert
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 1/9 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wedge Insert (N=9) | Flat Insert (N=3)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient experienced increased pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT02254473/Prot_SAP_000.pdf